CLINICAL TRIAL: NCT02853500
Title: Effect of Surefire Infusion Device on Tumor Response to Regional Intra-arterial Therapy for Primary Liver Malignancies
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled. Inability to perform intraprocedural MRI with the intraarterial infusion catheter in place due to MRI incompatibility.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Dmitry Rabkin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-077
Record Dates: First submitted 2016-06-30; First posted 2016-08-03 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Liver Cancer
Keywords: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TACE Procedure With TriNav (Experimental): Patients will receive a single administration of intra-arterial chemotherapy (Doxorubicin) during the TACE procedure via TriNav.
  * Patients will undergo structural follow-up for a timeframe of one year post treatment
  * Post-procedural, contrast-enhanced Magnetic Resonance Imaging (MRI) will be performed one month after trial entry, and at regular intervals thereafter for a total of one year to assess tumor response
  Interventions: Device: TriNav; Drug: Doxorubicin
- TACE Procedure Traditional Delivery (Active Comparator): Patients will receive a single administration of intra-arterial chemotherapy (Doxorubicin) during the TACE procedure via Traditional Delivery.
  * Patients will undergo structural follow-up for a timeframe of one year post treatment
  * Post-procedural, contrast-enhanced Magnetic Resonance Imaging (MRI) will be performed one month after trial entry, and at regular intervals thereafter for a total of one year to assess tumor response
  Interventions: Device: Traditional Delivery; Drug: Doxorubicin

INTERVENTIONS:
Device: TriNav — TriNav is a modified microcatheter with an expandable cone at its tip to prevent retrograde reflux of flow and change flow dynamics downstream.
  Arms: TACE Procedure With TriNav
Device: Traditional Delivery — Low profile tubing microcatheter for easier access to more peripheral/distal vascular branches for precise targeted delivery of medications.
  Arms: TACE Procedure Traditional Delivery
Drug: Doxorubicin — Medication used in cancer chemotherapy, including intraarterial delivery for liver malignancies.
  Other Names: Adriamycin

SUMMARY:
This research study is studying the TriNav ("TriSalus") for increasing delivery of chemotherapeutic agents delivered trans-arterially to intermediate stage Hepatocellular Carcinoma ("HCC") (Barcelona Clinic Liver Cancer (BCLC) class B; locally advanced, liver restricted disease patients.

The names of the study interventions involved in this study are:

-Trans-arterial chemoembolization ("TACE") with or without the utilization of Surefire

DETAILED DESCRIPTION:
This research study is a randomized Pilot study, which is the first time investigators are examining use of the TriNav device to improve tumor perfusion. Specifically, this study compares TACE both with or without the use of the TriNav device

Investigators are doing this research to determine if a TriNav Infusion System can improve tumor response to liver-directed intra-arterial chemotherapy compared to a traditional microcatheter.

TriNav is a Food and Drug Administration-approved valve-like device that blocks backflow within the artery but also generates increased pressure in a tumor feeder vessel during infusion. During this study, participants will receive the same medication in the same dose and the same way it would be delivered to the liver as a standard of care procedure, only either through a regular microcatheter (which is the standard of care procedure) or a TriNav Infusion System (which is a modified microcatheter).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable HCC, defined by imaging criteria or cytohistologic assessment. TACE as a preferred method of treatment is determined by a multidisciplinary Brigham and Women's Hospital / Dana Farber Cancer Institute (BWH/DFCI) Liver Tumor Board.
* Intermediate stage HCC (BCLC class B), not eligible for curative treatment, but with Child-Pugh A or B. Additionally, tumor cannot involve greater than 50% of the entire liver.
* Prior systemic chemotherapy is allowable.
* Age 18-75 years. The pediatrics population is not included as this disease has very low prevalence in that population.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Life expectancy of greater than at least 12 months.
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥60,000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate Aminotransferase (AST)/Alanine Aminotransferase (ALT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits or,
  * creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* No previous regional treatment (includes surgery, radiation or liver-directed arterial or ablative therapy).
* Main tumor size > 1 cm
* The effects of the study arm on the developing human fetus are unknown, however they are no different than for those in the control group. In addition, because significant radiation will be delivered during the procedure, a positive pregnancy test will exclude patients from the study in addition to excluding them from receiving standard therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had prior local regional therapy including radiation therapy, trans-arterial therapy, or ablative therapy.
* A hypovascular tumor (defined as a tumor with all its parts less contrast-enhanced than the non-tumorous liver parenchyma on arterial phase computed tomography scans).
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Evidence of hepatic decompensation including esophageal or gastric variceal bleeding or hepatic encephalopathy.
* Severe underlying cardiac or renal diseases.
* Color Doppler ultrasonography showing portal vein tumor thrombosis with complete main portal vein obstruction without cavernous transformation; or obstructive jaundice.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human Immunodeficiency Virus (HIV)-positive patients are NOT excluded from the study.
* Patients who cannot undergo MRI evaluation/examination (eg. pacemaker or other metallic implant)
* History of allergic reactions attributed to agents used in study (i.e. doxorubicin, epirubicin, MRI contrast agents or iodinated contrast agents).
* Pregnant women are excluded from this study because the chemotherapy utilized within the chemoembolic agent is teratogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemoembolic agent, breastfeeding should be discontinued if the mother is treated with chemoembolic agent. These potential risks may also apply to other agents used in this study as well as from the radiation associated with the angiographic procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Capillary permeability (Ktrans) calculated by software that analyzes enhancement on post-contrast MRI. | 2 years
  Ktrans represents a calculated metric that represents a measure of capillary permeability obtained during dynamic contrast enhanced MRI; it represents an absolute value of tracer concentration within the tissue of interest. It is calculated by measuring the accumulation of contrast agent on post-contrast MR images within a given tissue over time and comparing it to a baseline contrast-filled structure such as a blood vessel. The measurement represents accumulation of contrast for a given tissue, as determined by the investigator.
  Normality of the distribution will be tested using Shapiro-Wilk test. To compare Ktrans, the investigators will apply t-test or Wilcoxon rank sum test as appropriate.

SECONDARY OUTCOMES:
Extravascular extracellular volume fraction (ve) calculated by software that analyzes enhancement on post-contrast MRI. | 2 years
  Calculation of this value allows for more detailed analysis of contrast-enhancement of the tissue of interest. It represents an absolute value of tracer concentration within the tissue of interest, similar to Ktrans.
Rate constant (kep) | 2 years
  Calculation of this value allows for more detailed analysis of contrast-enhancement of the tissue of interest. It represents a derived value (kep = ktrans/ve) and is dependent upon ktrans and ve.
Plasma volume (vp) calculated by software that analyzes enhancement on post-contrast MRI. | 2 years
  Calculation of this value allows for more detailed analysis of contrast-enhancement of the tissue of interest. It represents an absolute value of tracer concentration within the plasma and allows for more accurate measurement of tissue permeability.
Time To Tumor Progression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Rabkin, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No